CLINICAL TRIAL: NCT04880668
Title: Impact of Aerosol Box Use on Patterns of Healthcare Provider and Environmental Contamination During Aerosol Generating Medical Procedures: A Multicenter Study
Brief Title: Impact of Aerosol Box Use on Healthcare Provider Contamination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KidSIM Simulation Program (Network)
Collaborators: International Network for Simulation-based Pediatric Innovation, Research and Education (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REB20-0893
Record Dates: First submitted 2021-04-27; First posted 2021-05-11 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Coronavirus; Covid19; COVID-19 Acute Respiratory Distress Syndrome
Keywords: simulation; AGMP; aerosol generating medical procedure; intubation; bag valve mask ventilation; laryngeal mask airway
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, two study arms
Masking Description: Unable to blind due to the nature of the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - No aerosol box (No Intervention): Participants will perform the AGMP without an aerosol box
- Intervention - Aerosol box (Experimental): Participants will perform the AGMP with an aerosol box
  Interventions: Device: Aerosol Box (Splashguard)

INTERVENTIONS:
Device: Aerosol Box (Splashguard) — The aerosol box is a transparent, plastic cube covering the patient's head and shoulders, with circular access ports on the front of the box allowing for access to manage the airway. An additional four access holes (i.e. two on either side of the box) allow for airway assistants to access the patient airway.
  Arms: Intervention - Aerosol box

SUMMARY:
Aerosol Generating Medical Procedures (AGMP) are procedures that have the potential to create tiny particles suspended in the air. These particles can contain germs such as viruses. The current Coronavirus Disease 2019 (COVID-19) pandemic is caused by the novel severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Patients infected with SARS-CoV-2 experience unusually high rates of critical illness that needs advanced airway management and intensive care unit admission. Bag-valve-mask (BVM) ventilation, laryngeal mask airway insertion (LMA), and endotracheal Intubation (ETI) are common AGMP for critically ill COVID-19 patients, and may contribute to a high risk of infection amongst Health Care Workers (HCW). To lessen HCW risk during high-risk AGMPs, a device called an aerosol box has been developed to place over the head of the patient, shielding the provider's face from virus droplets suspended in the air.

The purpose of this research study is to better understand how particles disperse during AGMPs. The project team hopes what is learned from the project can help inform infection control measures. This could help make changes to the clinical environment and make it safer for HCW's. The investigators intend to investigate how an aerosol box performs in reducing contamination of HCW's who perform critical airway interventions.

DETAILED DESCRIPTION:
The investigators plan to conduct a prospective, randomized controlled trial at four INSPIRE network sites (Alberta Children's Hospital, Ste. Justine Hospital, and Children's Hospital of Los Angeles and The Hospital for Sick Children). Simulation-based research confers the advantage of answering research questions without risk of harm to HCPs or patients, which is particularly important when studying a disease process with high mortality. Ethics approval has been submitted at all sites. Two participants will form an airway team, recruited to play the roles of airway provider and airway assistant for management of a simulated, critically ill COVID-19 patient. Participants will be randomized by team into either the control arm (i.e. no aerosol box) or the intervention arm (i.e. use of aerosol box). Following randomization, all participants will view a short video orienting them to the simulated clinical environment. Intervention arm teams will view an additional 5-minute video orienting them to the use of the aerosol box, and receive up to 15 minutes of hands-on training (see below for details). After orientation, teams will participate in three sequential simulation scenarios. The order of scenario delivery will be randomized to eliminate scenario order as a potential confounder. The location and nature of equipment, temperature and humidity within the resuscitation room will be standardized across all sites. A Laerdal Resusci-Anne manikin will be used as a simulated patient.

The aerosol box is a transparent, plastic cube covering the patient's head and shoulders, with circular access ports on the front of the box allowing for access to manage the airway. An additional four access holes (i.e. two on either side of the box) allow for airway assistants to access the patient airway. As our study includes only one airway assistant, the two holes that are not in use will be sealed shut during the study. The airway assistant will be directed to stand in a standardized position, to the immediate right of the airway provider. In a prior study, an aerosol box placed over the head of an adult volunteer demonstrated air leaks out of the box during exhalation and coughing that could be eliminated with the addition of a plastic drape. For this reason, the investigators have incorporated a plastic drape extending from the top of the box down to the patient's chest to prevent spread of aerosols. In another experiment, the addition of continuous wall suction to the aerosol box setup resulted in significantly decreased airborne particle exposure (for the airway provider) compared to aerosol box use without suction. Given that wall suction is ready available and accessible in most acute care areas, the aerosol box setup will include wall suction, with suction tubing running into the aerosol box at one point along the bottom of the box near the head of the patient. Wall suction will be set at 200 mmHg, which is consistent with the pressure used in prior studies to generate a negative airflow of approximately 50 L/min.

All participants (i.e. airway provider and airway assistant) randomized to the intervention arm will receive aerosol box training. A 5-minute video will orient participants to the design of the aerosol box and include expert-modeled demonstration of strategies for optimal BVM ventilation, ETI, and LMA insertion using an aerosol box with a 2-person airway team. The training video will be shot in English and French to permit viewing across study sites in Alberta, Ontario and Quebec. After viewing the video, participants will work in pairs to practice all three procedures for a maximum of 15 minutes, providing them opportunity to coordinate their movements to optimize efficiency. After each procedure, the participants will receive feedback from a local airway and aerosol box expert (i.e. site investigator).

The amount of aersolization that occurs in real patients is highly variable and dependent upon many factors (e.g. viral load, method of aerosolization, etc.), making it impossible to exactly replicate aerosolization of SARS-CoV-2 virus in the simulated environment. In this study, the investigators aim to create a model of aerosolization by standardizing various aspects of care (e.g. ventilation pressures, particle size and volume deposited, lung compliance), thus allowing us to make comparisons between different contexts (ie. aerosol box vs no box; BVM vs. LMA vs. ETI). To visualize aerosolization of particles, the study team will adapt methodology successfully utilized in studies evaluating aerosolization during airway management. GloGerm©™(Glo Germ Company, Moab, UT, USA) is a nontoxic, invisible fluorescent resin marker that illuminates when exposed to ultraviolet (UV) light. The SARS-CoV-2 virus requires a water and mucus envelope to spread, with the size of these virus-containing envelopes varying from larger droplets (>60 µm) to smaller airborne particles or infectious droplet nuclei (5-10 µm diameter). With a particle size of approximately 5 µm, Glo Germ™ represents a reasonable surrogate for aerosolized SARS-CoV-2. AGMPs can generate aerosols in two ways: by mechanically inducing and dispersing aerosols, or by inducing the patient to cough to produce aerosols. This study focuses on aerosols mechanically induced by three commonly performed AGMPs: BVM ventilation, LMA insertion, and ETI. Glo Germ™(0.5 mL) will be applied to the oropharynx and trachea of the manikin to simulate secretions. Glo Germ™ will be aerosolized from the mechanical pressures and airflow associated with bagging, or from manipulation of the airway, which is consistent with the current understanding of aerosolization mechanics in AGMPs. Participants will titrate ventilation pressures to 20 cm H2O peak inspiratory pressure, and 5-6 cm H2O peak end expiratory pressure using a digital pressure manometer that provides real-time feedback. Pilot work done using the methods (and ventilation pressures) described above resulted in contamination on the hands, torso, face shield, and feet of airway providers during BVM ventilation. This suggests these methods are sufficient to produce a measurable amount of Glo Germ™ particles during manual ventilation.

Prior to each scenario, all participants will donn personal protective equipment (PPE), consisting of: a gown, nitrile gloves, face shield, googles, and a N95 respirator. The brand, type and size of gowns and face shields will be standardized across all sites. PPE will be donned with a partner, guided by a standardized PPE donning checklist, and checked by a research assistant prior to the scenarios. All scenarios are 5 minutes in duration and tightly standardized by using a scenario template with pre-scripted patient progression. Intervention arm teams will use the aerosol box in all three scenarios while control arm teams will not use the aerosol box. At the end of the entire session, participants will receive an educational debriefing to discuss performance issues, infection control measures, and technical skills using a blended-method approach to debriefing. Doffing will occur in conjunction with a PPE partner, and guided by a standardized PPE doffing checklist to ensure consistency.

Scenario A: BVM Ventilation - depicts an adolescent patient with suspected COVID-19, presenting with progressive respiratory distress and desaturation. Participants will be directed to initiate BVM ventilation with a HEPA filter as per guidelines for managing COVID-19 pediatric patients. Aerosolization of particles occurs during manual ventilation, while the mask is on the patient's face. The scenario will last a total of 5 minutes.

Scenario B: ETI - depicts an adult patient with suspected COVID-19, presenting with progressive respiratory failure requiring intubation. In this scenario, providers will be advised by the team leader not to initiate BVM ventilation, which is consistent with AHA guidelines for adult COVID-19 patients requiring airway management. Participants will be directed to sedate, paralyze and intubate the patient using a videolaryngoscope (e.g. GlideScopeTM), and provide manual ventilation after intubation with a HEPA filter in place. The scenario will last a maximum of 5 minutes, or until the patient is successfully intubated, whichever is longer.

Scenario C: LMA Insertion - depicts the same patient as in Scenario B. In this scenario, providers will be advised by the team leader to insert an LMA. Participants will be directed to sedate, paralyze and intubate the patient, and provide manual ventilation after LMA insertion with a HEPA filter in place. The scenario will last a maximum of 5 minutes, or until the patient is successfully intubated, whichever is longer.

Data collection will occur immediately after each scenario, prior to and after doffing of PPE (see outcomes below). After data collection, the resuscitation room and airway trainer will be cleaned. Clean PPE will be provided for all participants for each scenario. These measures will ensure there is no incremental accumulation of GloGermTM particles from prior scenarios. All scenarios will be videotaped from a birds-eye view angle at the head of the bed. Video from the video laryngoscopy device will be captured during Scenario B.

Randomization will occur at the level of the team, stratified by study site and sex of the airway provider (to ensure equal distribution of sex in both arms), and conducted in blocks of 4 to ensure an even distribution of teams across study arms. Randomization packages will be prepared at a central study side using a web-based random number generator. Sequentially numbered recruitment packages provided for each site will contain sealed opaque envelopes (i.e. one envelope per study arm) with study arm assignments and unique identifier codes for participants.

Sample size estimation is based on primary outcome measure. Given the paucity of quantitative research in this area, the investigators propose a sample of 60 teams (120 participants) in total, or 30 teams (60 participants) per study arm. As each team will receive repeated measures (i.e. 3 scenarios), this sample size permits detection of a medium effect size (Cohen's d = 0.65), with a significance level of 0.05, a power of 0.8, and a high intra-cluster correlation coefficient (rho = 0.7) to make a conservative estimation. Accounting for missing data due to technical issues, the investigators will recruit one extra team per study group at each site. Therefore, the total sample size will be 66 teams (132 participants).

ELIGIBILITY:
Inclusion Criteria (Airway Provider):

* Healthcare provider from inpatient unit, intensive care unit, operating room unit and/or emergency department
* Attending physician or fellow in emergency medicine, intensive care, pediatrics, or anesthesia
* Adult or Pediatric Advanced Life Support certification

Inclusion Criteria (Airway Assistant)

* Healthcare provider from inpatient unit, intensive care unit, operating room unit and/or emergency department
* Attending physician, resident, fellow, nurse or respiratory therapist
* Adult or Pediatric Advanced Life Support certification.

Exclusion Criteria:

* Decline to provide informed consent
* Unable to perform tasks required of the role due to physical limitations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All genders eligible
Enrollment: 122 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Change in Integrated Density (Pre vs Post Doffing) | Immediately after each procedure (BVM, ETI, LMA)
  Integrated density of HCP contamination, quantified from digital photos of GloGerm™ deposited on the airway team members pre and post-doffing.
Change in Area of contamination (Pre vs Post Doffing) | Immediately after each procedure (BVM, ETI, LMA)
  Quantified from digital photos of GloGerm™ deposited on the airway team members pre and post-doffing.

SECONDARY OUTCOMES:
Time to task completion | Immediately after ETI and LMA procedures
  time to successful intubation or LMA insertion (captured by video review by 2 trained and calibrated raters)
First pass success rate | Immediately after ETI and LMA procedures
  first pass success rate for ETI and LMA insertion (captured by video review by 2 trained and calibrated raters)
Number of healthcare providers contaminated | Immediately after each procedure (BVM, ETI, LMA)
  Number of healthcare providers contaminated
Number of different body parts contaminated | Immediately after each procedure (BVM, ETI, LMA)
  Number of different body parts contaminated
Environmental Contamination | Immediately after each procedure (BVM, ETI, LMA)
  integrated density of environmental contamination, captured by taking a photo of the room in standardized conditions
Provider Workload | Immediately after each procedure (BVM, ETI, LMA)
  Provider workload as measured by NASA TLX survey, rated on a scale of 0-20, with 20 being maximum workload for each element
Quality of intubation performance | Immediately after ETI
  Quality of intubation performance (captured by video review of both video laryngoscopy and video from within the room) assessed using a previously published intubation checklist; rated on a scale of 0 to 41, with 41 being perfect performance
Provider opinions on aerosol box | Immediately after all 3 procedures are completed
  pros and cons of using aerosol box, captured by questionnaire completed by both participants (multiple choice and open field question types)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Cheng, MD, Principal Investigator — University of Calgary
Locations (4):
- Department of Emergency Medicine, Children's Hospital of Los Angeles, Los Angeles, California, United States
- Canada (3):
  - KidSIM-ASPIRE Simulation Research Program Alberta Children's Hospital, Calgary, Alberta
  - Department of Pediatrics, The Hospital for Sick Children, Toronto, Ontario
  - Department of Pediatrics, CHU Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No
No plan to share data with other researcher. Potential sharing may be possible upon individual request with justification.

REFERENCES:
- [Derived] Cheng A, Pirie J, Lin Y, Lo CY, Davidson J, Chang T, Matava C, Buyck M, Harel DS, Collia N, Neveu G, Pellerin S, Madadi M, Manshadi K, Wan B, Levy A; International Network for Simulation-based Pediatric Innovation, Research and Education (INSPIRE) Aerosol-Generating Medical Procedure (AGMP) Investigators. Aerosol Box Use in Reducing Health Care Worker Contamination During Airway Procedures (AIRWAY Study): A Simulation-Based Randomized Clinical Trial. JAMA Netw Open. 2023 Apr 3;6(4):e237894. doi: 10.1001/jamanetworkopen.2023.7894. PMID 37043197